CLINICAL TRIAL: NCT04837183
Title: Catheter Ablation of Ventricular Arrhythmia Reduces Skin Sympathetic Activity
Status: Terminated | Type: Observational
Why Stopped: This study was closed before its planned primary completion date because early data indicated that VT ablation had little impact on sympathetic nerve activity in short-term follow up.
Sponsor: Mayo Clinic (Other)
Collaborators: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Yong-Mei Cha, Principal Investigator, Mayo Clinic
Other Study IDs: 20-001448
Record Dates: First submitted 2021-03-16; First posted 2021-04-08 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being done to determine whether there is an increase in sympathetic nerve activity before the onset of ventricular arrhythmias or irregular heartbeat rhythm. In addition, this study is looking at the relationship between sympathetic nerve activity and how patients with ventricular arrhythmias respond to catheter ablation treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have non-sustained or sustained VA (VA ≥ 30s or receiving appropriate ICD therapies) are presented to the clinic or admitted to the hospital within 7 days of episodes.
* The causes of VA are associated with structural heart diseases including ischemic or nonischemic cardiomyopathy (idiopathic cardiomyopathy, hypertrophic cardiomyopathy, cardiac sarcoidosis or amyloidosis, and arrhythmogentic right ventricular dysplasia).
* Subjects are 18 years of age and older.

Exclusion Criteria:

* Female patients who is pregnant or of childbearing potential and not on a reliable form of birth control.
* Allergic to skin patch electrodes.
* Vulnerable populations (fetuses, neonates, pregnant women, prisoners, institutionalized individuals).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients will undergo catheter ablation to control VA recommended by current guideline.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in amplitude of skin sympathetic nerve activity | Baseline, 24 hours post catheter ablation and approximately 3-6 months post-operative
  measured in µV
Change in LF/HF ratio | Baseline, 24 hours post catheter ablation and approximately 3-6 months post-operative
  low frequency (LF)/high frequency (HF) ratio of the skin sympathetic nerve activity

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Mei Cha, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials